CLINICAL TRIAL: NCT00199186
Title: A Randomized, Multicenter Open Label Phase II Study to Determine the Safety and Efficacy of Induction Therapy With Imatinib in Comparison With Standard Induction Chemotherapy in Elderly (> 55 Years) Patients With Ph Positive Acute Lymphoblastic Leukemia (ALL)
Brief Title: Study Comparing Imatinib With Chemotherapy as Induction in Elderly Patients With Philadelphia Positive Acute Lymphoblastic Leukemia (ALL)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSTI571ADE10; GMALL-STI571-ELDERLY-01/02
Record Dates: First submitted 2005-09-16; First posted 2005-09-20 (Estimated); Last update posted 2007-10-19 (Estimated); Status verified 2005-09

CONDITIONS: Philadelphia Positive Acute Lymphoblastic Leukemia; Lymphoid Blastic Phase of Chronic Myeloid Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Imatinib Mesylate; Vincristine; Cyclophosphamide; Cytarabine; Dexamethasone; Idarubicin; Methotrexate

INTERVENTIONS:
Drug: imatinib
Drug: vincristine
Drug: cyclophosphamide
Drug: cytosine arabinoside
Drug: dexamethasone
Drug: idarubicin
Drug: methotrexate (intrathecal)
Drug: AraC (intrathecal)
Drug: dexamethasone (intrathecal)

SUMMARY:
The aims of the study are to determine whether single agent imatinib (STI571; Glivec) is more effective as up-front remission induction therapy than conventional multi-agent induction chemotherapy for elderly patients with Philadelphia positive (Ph+)ALL, whether this treatment is better tolerated, and whether subsequent combination therapy with imatinib and chemotherapy of approximately a 1 year duration is tolerable and effective with respect to maintaining remissions.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients
* Age > 55 years (biological age)
* Diagnosis of Ph1 chromosome-positive ALL (pre-B, common- or pre-pre-B ALL)
* Newly diagnosed, lymphoid blast crisis of chronic myeloid leukemia
* Only pre-phase chemotherapy prior to study start
* World Health Organization (WHO) status 0, 1 or 2
* Voluntary written informed consent

Exclusion Criteria:

* Creatinine levels more than 2 x the upper limit of normal (ULN)
* Total serum bilirubin more than 1.5 x the ULN
* AST (SGOT) or ALT (SGPT) more than 5 x the ULN
* Any other prior antineoplastic treatment except for pre-phase chemotherapy
* Active central nervous system (CNS) leukemia
* New York Heart Association (NYHA) grade 3/4 cardiac disease
* Active severe infection
* Serious concomitant medical condition
* Patients with a history of non-compliance to medical regimens

Min Age: 56 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-03

PRIMARY OUTCOMES:
Remission rate after induction therapy

SECONDARY OUTCOMES:
Mortality rate during induction
Severe adverse events during induction
Efficacy of salvage therapy after crossover
Levels of minimal residual disease
Incidence of relapse
Remission duration
Disease free survival
Overall survival
Frequency of point mutations in the BCR-ABL gene

CONTACTS AND LOCATIONS:
Overall Officials: Oliver G Ottmann, M.D., Study Chair — Medizinische Klinik II, Johann Wolfgang Goethe Universität
Locations (1):
- Medizinische Klinik II, Johann Wolfgang Goethe Universität, Frankfurt am Main, Germany